CLINICAL TRIAL: NCT07404761
Title: A Multicenter, Randomized, Controlled Study to Evaluate the Efficacy and Safety of the SSMD in Neuromotor Rehabilitation
Brief Title: Safety and Effectiveness of Spatial StimelMD (SSMD) in Subjects With Upper Limb Neuromotor Impairments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Motion Informatics LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-SSMD-01
Record Dates: First submitted 2026-02-02; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Stroke; Upper-limb Motor Impairment; Hemiparesis; Spinal Cord Injury; Traumatic Brain Injury
Keywords: randomized; ssmd; neuromotor rehabilitation
MeSH Terms: conditions — Stroke; Paresis; Spinal Cord Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Participants are randomized into two parallel groups to receive either SSMD therapy plus standard rehabilitation care or standard functional electrical stimulation (FES) plus standard care over approximately 5-6 weeks.
Masking Description: Not applicable. This is an open-label study with no masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- SSMD Therapy + Standard Care (Experimental): Participants receive Spatial StimelMD (SSMD) therapy in addition to standard rehabilitation care. Treatment includes approximately 25 supervised sessions delivered over 5-6 weeks.
  Interventions: Device: Spatial StimelMD (SSMD)
- Standard FES + Standard Care (Active Comparator): Participants receive standard functional electrical stimulation (FES) in addition to standard rehabilitation care. Treatment includes approximately 25 supervised sessions delivered over 5-6 weeks.
  Interventions: Device: Functional Electrical Stimulation (FES)

INTERVENTIONS:
Device: Spatial StimelMD (SSMD) — Spatial StimelMD (SSMD) is a device-based neuromotor rehabilitation intervention used for upper-limb therapy. Participants receive SSMD therapy in supervised sessions as part of a structured rehabilitation program over approximately 5-6 weeks (about 25 sessions).
  Arms: SSMD Therapy + Standard Care
Device: Functional Electrical Stimulation (FES) — Functional electrical stimulation (FES) is a standard device-based intervention used in rehabilitation to stimulate muscle activation for upper-limb therapy. Participants receive FES in supervised sessions as part of standard rehabilitation care over approximately 5-6 weeks (about 25 sessions).
  Arms: Standard FES + Standard Care

SUMMARY:
This is a multicenter, randomized, controlled clinical study evaluating the safety and effectiveness of the Spatial StimelMD (SSMD) device for upper-limb neuromotor rehabilitation in adults with impairment following stroke or traumatic brain injury (TBI).

Participants will be randomized to receive either SSMD therapy plus standard rehabilitation care or standard functional electrical stimulation (FES) plus standard care. Subjects will complete approximately 25 supervised treatment sessions over 5-6 weeks, with assessments at baseline, mid-treatment, post-treatment (primary endpoint), and a 1-month follow-up.

The primary effectiveness endpoint is improvement in upper-limb motor function measured by the Fugl-Meyer Upper Extremity (FMA-UE) assessment. Secondary outcomes include movement metrics, EMG signal strength, functional independence, usability measures, and adverse event monitoring.

The study plans to enroll approximately 150 subjects to achieve 126 completers, across 2-6 clinical sites.

DETAILED DESCRIPTION:
CP-SSMD-01 is a multicenter, randomized, controlled clinical study designed to evaluate the safety and effectiveness of the Spatial StimelMD (SSMD) device for upper-limb neuromotor rehabilitation in adults with impairment following stroke or traumatic brain injury (TBI). The study compares SSMD therapy plus standard rehabilitation care to standard functional electrical stimulation (FES) plus standard care. Participants will complete approximately 25 supervised treatment sessions over a 5-6 week period.

Subjects will undergo evaluations at baseline, mid-treatment, post-treatment (the primary endpoint), and a follow-up visit approximately one month after completing therapy. The primary outcome measure is improvement in upper-limb motor function assessed using the Fugl-Meyer Assessment for the Upper Extremity (FMA-UE). Secondary outcomes include additional measures of motor performance and movement quality, EMG-based muscle activation metrics, functional independence outcomes, usability assessments, and safety monitoring through adverse event reporting.

The study aims to enroll approximately 150 participants, with an expected 126 completing the full protocol, across 2-6 clinical sites. This trial is intended to generate clinical evidence on whether SSMD therapy can support meaningful upper-limb motor recovery compared with a standard stimulation-based rehabilitation approach in individuals affected by stroke or TBI.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-80 years.
2. Clinically confirmed diagnosis of stroke or TBI within the past 12 months.
3. Presence of moderate to severe neuromotor impairment in at least one limb, as evidenced by medical evaluation and a score <35 on the Fugl-Meyer Upper Extremity motor subscale (FMA-UE).
4. Capacity and willingness to provide informed consent, indicating understanding of the study purpose, procedures, and potential risks and benefits.
5. Subject is able to adhere to the study schedule and cognitively capable to perform the treatment.
6. Stable medical condition without ongoing acute complications that could interfere with participation.

Exclusion Criteria:

1. Presence of contraindications to electrical stimulation (ES), including implanted electronic medical devices (e.g., pacemakers, insulin pumps) or conditions that may be exacerbated by electrical stimulation (e.g., uncontrolled epilepsy).
2. Individuals with medical conditions, which are prone to seizures or motion sensitivity, at the investigator's discretion.
3. Individuals with light sensitivity, as the AR component may involve visual stimuli that could cause discomfort or adverse reactions in these patients.
4. Individuals with acute physical conditions or injuries that could interfere with the proper placement of the electrodes or safe use of the device.
5. Presence of spinal shock or unresolved acute spinal cord dysfunction, characterized by complete loss of reflexes, flaccid paralysis, or autonomic instability.
6. Current participation in other clinical trials that could confound the study results.
7. Severe cognitive impairment that precludes the ability to provide informed consent or reliably adhere to the study protocol, as determined by cognitive screening and clinical judgment.
8. Women who are pregnant, nursing, or who plan to become pregnant while in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment - Upper Extremity (FMA-UE) | Baseline to end of treatment (post-treatment; approximately 5-6 weeks)
  Change from baseline to end of treatment in the Fugl-Meyer Assessment Upper Extremity (FMA-UE) motor function score (range 0-66), with higher scores indicating better motor function (better outcome).

SECONDARY OUTCOMES:
Movement Quality (SSMD Assessment Mode) | Baseline to end of treatment (approximately 5-6 weeks)
  Change in upper-limb movement quality measured using SSMD assessment mode metrics.
EMG Signal Strength (Threshold) | Baseline to end of treatment (approximately 5-6 weeks)
  Change in EMG signal strength (threshold) measured during study assessments.
Functional Independence Measure (FIM) | Baseline to end of treatment (approximately 5-6 weeks)
  Change from baseline to end of treatment in the Functional Independence Measure (FIM) total score (range 18-126), with higher scores indicating greater functional independence (better outcome).

OTHER OUTCOMES:
Modified Ashworth Scale (MAS) | Baseline to end of treatment (approximately 5-6 weeks)
  Change from baseline in spasticity measured by the Modified Ashworth Scale (range 0-4; higher scores indicate worse spasticity).
  Time Frame: Baseline to end of treatment (5-6 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Boris Chelibian, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.